CLINICAL TRIAL: NCT01131195
Title: Safety and Tolerability of Bevacizumab Plus Paclitaxel vs. Bevacizumab Plus Metronomic Cyclophosphamide and Capecitabine as First-Line Therapy in Patients With HER2-Negative Metastatic or Locally Recurrent Breast Cancer - A Multicenter, Randomized Phase III Trial.
Brief Title: Metronomic Therapy in Metastatic Breast Cancer.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 24/09; SWS-SAKK-24-09; EU-21025; CDR0000669252
Record Dates: First submitted 2010-05-25; First posted 2010-05-26 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Breast Cancer
Keywords: HER2-negative breast cancer; recurrent breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Paclitaxel; Cyclophosphamide; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A: bevacizumab and paclitaxel (Active Comparator): Bevacizumab (10 mg/kg) i.v. is given every two weeks. Paclitaxel (90 mg/m2) i.v. is given on days 1, 8, and 15 of a 4 week cycle. Both medications are given until PD, unacceptable adverse event, or consent withdrawal. If an unacceptable adverse event to any of the drugs in this treatment arm occurs the remaining tolerated drug is given until PD, consent withdrawal, or unacceptable adverse event according to local investigators opinion.
  Interventions: Biological: bevacizumab, Paclitaxel
- Arm B: bevacizumab, cyclophosphamide and capecitabine (Active Comparator): Bevacizumab (10 mg/kg) i.v. is given every two weeks. Cyclophosphamide (50 mg) and capecitabine (3x 500 mg) p.o. are given daily. All three medications are given until PD, unacceptable adverse event, or consent withdrawal. If an unacceptable adverse event to any of the drugs in this treatment arm occurs the remaining tolerated drug(s) is (are) given until PD, consent withdrawal, or unacceptable adverse event according to local investigators opinion
  Interventions: Biological: Bevacizumab, Cyclophosphamide, Capecitabine

INTERVENTIONS:
Biological: bevacizumab, Paclitaxel — Bevacizumab (10 mg/kg) i.v. is given every two weeks. Paclitaxel (90 mg/m2) i.v. is given on days 1, 8, and 15 of a 4 week cycle.
  Other Names: Avastin
  Arms: Arm A: bevacizumab and paclitaxel
Biological: Bevacizumab, Cyclophosphamide, Capecitabine — Bevacizumab (10 mg/kg) i.v. is given every two weeks. Cyclophosphamide (50 mg) and capecitabine (3x 500 mg) p.o. are given daily
  Other Names: Avastin; Xeloda
  Arms: Arm B: bevacizumab, cyclophosphamide and capecitabine

SUMMARY:
RATIONALE: Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Drugs used in chemotherapy, such as paclitaxel, cyclophosphamide, and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. It is not yet known whether bevacizumab is more effective when given together with paclitaxel or cyclophosphamide and capecitabine in treating patients with breast cancer.

PURPOSE: This randomized phase III trial is studying the side effects of giving bevacizumab together with paclitaxel and to see how well it works compared with giving bevacizumab together with cyclophosphamide and capecitabine as first-line therapy in treating women with locally advanced, recurrent, or metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine if bevacizumab and paclitaxel versus bevacizumab, metronomic cyclophosphamide, and capecitabine as first-line therapy causes less medication-related adverse events in women with HER2-negative metastatic, locally advanced, or recurrent breast cancer.
* To compare quality of life (QOL) in patients treated with these regimens.
* To replicate previous findings of better QOL in patients with complete response or partial response versus stable disease for 6 months or greater.
* To determine the predictive value of baseline QOL for the duration of a meaningful change in QOL of patients treated with chemotherapy.
* To determine the associations between the QOL endpoints, selected health economics, and clinical endpoints.

OUTLINE: This is a multicenter study. Patients are stratified according to tumor response (measurable vs evaluable disease), WHO performance status (0 or 1 vs 2), and center. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive bevacizumab IV over 30-90 minutes on days 1 and 15 and paclitaxel IV on days 1, 8, and 15. Treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive bevacizumab IV over 30-90 minutes on days 1 and 15, oral cyclophosphamide once daily on days 1-28, and oral capecitabine 3 times a day on days 1-28. Treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity.

Patients complete quality-of-life questionnaire (BL-QA) and health economics questionnaires (BL-HEA and EQ-5D) at baseline, during, and after completion of study therapy.

After completion of study treatment, patients are followed up at 1 month, every 3 months for 1 year, and then every 6 months for 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the breast

  * Locally advanced, recurrent, or metastatic disease
* HER2-negative disease
* Measurable or evaluable disease
* Candidate for taxane-based chemotherapy
* No presence or history of CNS metastasis

  * Clinical suspicion of CNS metastasis must be confirmed by CT or MRI scan
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* WHO performance status 0-2
* Neutrophil count ≥ 1.5 x 10^9/L
* Platelet count ≥ 100 x 10^9/L
* Hemoglobin ≥ 80 g/L
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST ≤ 5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN (≤ 5 times ULN in case of liver metastases or ≤ 10 times ULN in case of bone metastases)
* Serum creatinine ≤ 1.5 times ULN
* Urine protein < 2+ by dipstick OR ≤ 1 g by 24-hour urine collection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 12 months after completion of study therapy
* Patients with INR > 1.5 (or Quick ≤ 70%) OR aPTT > 1.5 times ULN within 7 days prior to expected first trial treatment must be receiving anticoagulant medication

  * Patients receiving full-dose oral or parental anticoagulants may be included in the trial provided anticoagulant dosing has been stable for at least 2 weeks prior to trial entry and the appropriate coagulation monitoring tests are within local therapeutic limits
* Must be compliant and geographically proximal for staging and follow-up
* No previous malignancy within the past 5 years except for adequately treated carcinoma in situ of the cervix or localized nonmelanoma skin cancer
* No known hypersensitivity to trial drugs or its active compound (e.g., fluoropyrimidine), any other components of the trial drugs, or drugs formulated with cremophor EL including hypersensitivity to Chinese hamster ovary cell products or any other humanized recombinant antibodies
* No preexisting peripheral motor or sensory neuropathy > NCI CTCAE grade 2 (i.e., moderate symptoms or limiting instrumental activities of daily living)
* No history or evidence of inherited bleeding diathesis, coagulopathy with the risk of bleeding, serious nonhealing wound, active peptic ulcer, nonhealing bone fracture, or bleeding metastases
* No history of abdominal fistula, grade 4 bowel obstruction, or gastrointestinal perforation or intra-abdominal abscess within the past 6 months
* No evidence of other medical conditions that would impair the ability of the patient to participate in the trial or might preclude therapy with trial drugs, including any of the following:

  * DPD deficiency
  * Severe respiratory, cardiac, hepatic, or renal disease
  * Active infection
  * Uncontrolled diabetes mellitus
  * Uncontrolled hypertension ≥ 140/100 mm Hg
  * Myocardial infarction within the past 12 months
  * Cerebrovascular accident or stroke within the past 6 months
  * History of hemorrhagic disorders
* No psychiatric disorder precluding understanding of information on trial-related topics, giving informed consent, filling out quality-of-life forms, or interfering with compliance for oral drug intake

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy for metastatic or locally recurrent breast cancer
* No prior radiotherapy for metastatic disease

  * Prior radiotherapy for the relief of metastatic bone pain allowed provided no more than 30% of marrow-bearing bone was irradiated
* At least 12 months since prior bevacizumab or other anti-VEGF therapy
* At least 12 months since prior capecitabine, continuous (> 24 hours) fluorouracil infusion, or other oral fluoropyrimidine (e.g., eniluracil/fluorouracil, uracil/tegafur, S1, or emitefur)
* At least 12 months since prior taxane-based chemotherapy
* At least 6 months since other prior (neo)adjuvant chemotherapy
* At least 30 days since prior treatment in another clinical trial
* At least 24 hours since prior minor surgical procedures
* At least 28 days since prior and no concurrent major surgical procedures (including open biopsy) and no anticipation of the need for major surgery during the first course of this trial
* At least 10 days since prior hormone therapy for metastatic disease
* No continuous daily treatment with corticosteroid except for inhaled steroids
* No concurrent chronic daily aspirin > 325 mg/day
* No concurrent chronic daily clopidogrel > 75 mg/day
* No other concurrent anticancer treatments
* No other concurrent investigational treatments or experimental drugs
* No other concurrent drug therapy contraindicated for use with the trial drugs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2010-07-19 (Actual); Primary Completion 2012-12-14 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Incidence of grade 3-5 adverse events | Documentation of AE observed during trial treatment and in follow-up until resolution
  Patients who have experienced at least one of the adverse event grade ≥ 3 according to the NCI CTCAE criteria 4.0 are considered for the primary endpoint.

SECONDARY OUTCOMES:
Objective response (OR) | the best response under trial treatment
  OR is the best response under trial treatment, defined as a complete response (CR) or partial response (PR) as assessed by RECIST v1.1.
Disease control (DC) | best response under trial treatment at 24 weeks after randomization
  DC is the best response under trial treatment, defined as CR + PR + stable disease.
Progression-free survival (PFS) | from randomization until documented tumor progression
  PFS is calculated from randomization until documented tumor progression according to RECIST 1.1 or death of any cause, whichever occurs first.
Overall survival (OS) | the time from randomization to death from any cause
  OS is defined as the time from randomization to death from any cause
Time to specific grade 3-5 adverse events | Time from randomization until the first occurrence of the predefined grade 3-5 adverse events for the primary endpoint.
  Time from randomization until the first occurrence of the predefined grade 3-5 adverse events for the primary endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Rochlitz, MD, Study Chair — Universitaetsspital-Basel; Ralph Winterhalder, MD, Study Chair — Luzerner Kantonsspital
Locations (23):
- Switzerland (23):
  - Hirslanden Klinik Aarau, Aarau
  - Kantonspital Aarau, Aarau
  - Kantonsspital Baden, Baden
  - Universitaetsspital-Basel, Basel
  - Spitalzentrum Biel, Biel
  - RSV-GNW Spitalzentrum Oberwallis, Brig
  - Kantonsspital Graubuenden, Chur
  - Kantonsspital Frauenfeld, Frauenfeld
  - Kantonsspital Freiburg, Fribourg
  - Hopital Cantonal Universitaire de Geneve, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital Luzern, Luzerne
  - Oncology Institute of Southern Switzerland - IOSI Ticino, Mendrisio
  - Kantonsspital Olten, Olten
  - Kantonsspital - St. Gallen, Sankt Gallen
  - Hopital Regional de Sion-Herens-Conthey, Sion
  - Regionalspital Thun, Thun
  - Spital Uster, Uster
  - Kantonsspital Winterthur, Winterthur
  - Onkozentrum - Klinik im Park, Zurich
  - Onkozentrum Hirslanden, Zurich
  - City Hospital Triemli, Zurich
  - UniversitaetsSpital Zuerich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rochlitz C, Bigler M, von Moos R, Bernhard J, Matter-Walstra K, Wicki A, Zaman K, Anchisi S, Kung M, Na KJ, Bartschi D, Borner M, Rordorf T, Rauch D, Muller A, Ruhstaller T, Vetter M, Trojan A, Hasler-Strub U, Cathomas R, Winterhalder R; Swiss Group for Clinical Cancer Research (SAKK). SAKK 24/09: safety and tolerability of bevacizumab plus paclitaxel vs. bevacizumab plus metronomic cyclophosphamide and capecitabine as first-line therapy in patients with HER2-negative advanced stage breast cancer - a multicenter, randomized phase III trial. BMC Cancer. 2016 Oct 10;16(1):780. doi: 10.1186/s12885-016-2823-y. PMID 27724870
- [Derived] Hoon SN, Lau PK, White AM, Bulsara MK, Banks PD, Redfern AD. Capecitabine for hormone receptor-positive versus hormone receptor-negative breast cancer. Cochrane Database Syst Rev. 2021 May 26;5(5):CD011220. doi: 10.1002/14651858.CD011220.pub2. PMID 34037241